CLINICAL TRIAL: NCT06069648
Title: Effects of Decision Aids on the Participation of South Asian Women in Cervical Cancer Screening: A Randomised Controlled Trial
Brief Title: Effects of Decision Aids on the Participation of South Asian Women in Cervical Cancer Screening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dorothy Ngo Sheung Chan, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HMRFSADA
Record Dates: First submitted 2023-09-22; First posted 2023-10-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; screening; South Asians; ethnic minority; decision aid
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Placebo Comparator): factsheet about healthy living
  Interventions: Behavioral: a leaftlet
- printed decision aid (Experimental): receive printed decision aid
  Interventions: Behavioral: printed screening decision aid
- mobile decision aid (Experimental): receive mobile decision aid
  Interventions: Behavioral: mobile screening decision aid

INTERVENTIONS:
Behavioral: printed screening decision aid — a booklet form of screening decision aid containing information of cervical cancer screening options
  Arms: printed decision aid
Behavioral: a leaftlet — a leaflet containing information about healthy lifestyles
  Arms: control
Behavioral: mobile screening decision aid — a mobile app format of screening decision aid containing information of cervical cancer screening options
  Arms: mobile decision aid

SUMMARY:
Objectives: To examine the effects of linguistically appropriate decision aids on decisional conflicts, risk perception, clarity of values, screening decisions and screening uptake among South Asian women in Hong Kong Design and subjects: A randomised controlled trial. A sample of 270 South Asian women aged 25-64 will be recruited to one of the two intervention groups or control group.

Instruments: A survey will be conducted to collect data on the variables of concern (decisional conflicts, risk perception, clarity of values, screening decision and screening uptake).

Interventions: Ethnically match community health workers (CHWs) will deliver the printed or mobile application decision aids to intervention group participants and briefly explain how to use the decision aid. The participants will choose a time and place of their convenience to read the decision aid. The participants will be contacted by CHWs within 2 weeks and asked if they have experienced any problems. Navigation assistance will be given as requested.

Main outcome measures: Decisional conflicts, risk perception, clarity of values, screening decision and uptake.

Data analysis: The repeated-measure outcomes of risk perception, clarity of values, decisional conflicts and screening decision will be compared between the three groups while adjusting for the stratifying variable (ethnicity) using a generalised estimating equation model, and a multivariable logistic regression with adjustment for ethnicity will be used to compare the screening uptake of the three groups.

Expected results: The decision aid will clarify the participants' values and help them to make screening decisions and increase the uptake.

ELIGIBILITY:
Inclusion Criteria:

1. Indian, Pakistani or Nepalese;
2. aged 25 to 64;
3. no history of cervical cancer or total hysterectomy;
4. have a history of sexual activity;
5. cannot understand Chinese but can read or communicate in English, Hindi, Urdu or Nepali;
6. have not had a Pap/HPV test in the past 3 years;
7. have and are willing to use a smartphone in this intervention.

Exclusion Criteria:

* NA

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 270 (Estimated)
Dates: Start 2024-07-11 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
decisional conflict | baseline and 2 weeks after intervention
  16-item Decisional Conflict Scale will be used to measure decisional conflict. The scale consists of five subscales: informed subscale, values clarity subscale, support subscale, uncertainty subscale and effective decision subscale. The scores will be converted to a 0-100 scale, giving a possible range of 0 (no decisional conflict) to 100 (extremely high decisional conflict). A score of 25 or below indicates that a person has low decisional conflict, and a score of 37.5 and above indicates that a person has decisional delay.
cervical cancer screening uptake | 3 months after intervention
  The participants will be asked 'Have you undergone cervical cancer screening in the past 3 months?

SECONDARY OUTCOMES:
risk perception | baseline and 2 weeks after intervention
  One question will be used to assess the participants' perceptions of their risk of cancer. Women will be asked to rate their risk of cervical cancer as low, moderate or high.
screening decision: choice predisposition | baseline and 2 weeks after intervention
  Choice predisposition assesses a person's leaning towards an option and is rated on a 15-point scale that ranges from 1 (leaning towards 'yes') to 15 (leaning towards 'no').
screening decision: choice question | baseline and 2 weeks after intervention
  The choice question asks about the screening decision and a question about the use of a screening option (Pap test/HPV testing). It is assessed using a 'no/yes/unsure' format.

IPD SHARING:
Plan to Share IPD: No